CLINICAL TRIAL: NCT04897074
Title: A Single Arm Pivotal Trial to Assess the Efficacy of AKL-T01, a Novel Digital Intervention Designed to Improve Attention, in Adolescents, Aged 13-17 Years Old, Diagnosed With Attention Deficit Hyperactive Disorder (ADHD)
Brief Title: Software Treatment for Actively Reducing Severity of ADHD in Adolescents (STARS-ADHD-Adolescents)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Akili-051
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AKL-T01 (Experimental): Digital Treatment
  Interventions: Device: AKL-T01

INTERVENTIONS:
Device: AKL-T01 — AKL-T01 multitasking digital treatment. AKL-T01 multitasking treatment employs perceptual discrimination attention/memory task as well as a continuous motor "driving" task.

SUMMARY:
The purpose of this study is to evaluate the effects of videogame-like digital therapy on attentional functioning and symptoms in adolescents ages 13-17 diagnosed with ADHD

DETAILED DESCRIPTION:
This study is a multi-center, unblinded/non-controlled study to evaluate objective attention functioning and ADHD symptoms and impairments in adolescents aged 13 to 17 years old, with a diagnosis of ADHD (combined or inattentive subtype), stably on or off ADHD medication, after 4-weeks of AKL-T01 treatment.

Up to 165 total participants from up to 20 sites will be enrolled.

During the Screening/baseline, participants will undergo screening to evaluate eligibility for the study. Eligible participants will continue onto baseline procedures in the same visit.

Treatment phase (Day 2-27) will involve using the digital therapy at home for each participant. Compliance with treatment/use requirements will be monitored remotely during this phase.

An In-Clinic assessment will be completed on Day 28 to assess key outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents between the ages of 13 and 17 years and 10 months at time of consent (must be under 18 years at study completion)
2. Confirmed diagnosis of ADHD combined or inattentive type, according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) as confirmed by MINI-Kid Version 7.0.2.
3. Stably on or off ADHD medication for ≥4 weeks prior to study enrollment and throughout the 4-week study
4. Baseline visit score on the TOVA-ACS score ≤ -1.8
5. Access to and self-report of ability to connect wireless devices to a functional wireless network
6. Ability to follow written and verbal instructions (English) as assessed by the PI and/or study coordinator
7. Able to comply with all testing and study requirements
8. Estimated IQ score ≥80 as assessed by the Kaufmann Brief Intelligence Test, Second Edition (KBIT-II)
9. Patient assent and caregiver informed consent
10. Stably on or off psychoactive medications for ≥4 weeks prior to study enrollment and throughout the 4-week study

Exclusion Criteria:

1. Current controlled or uncontrolled, comorbid psychiatric diagnosis that in the opinion of the Investigator may confound study data/assessments.
2. Participant is currently considered at risk for attempting suicide, has made a suicide attempt within the past year, or is currently demonstrating active suicidal ideation or self-injurious behavior, in the opinion of the Investigator based on the MINI-kid clinical interview.
3. Motor condition (e.g., physical deformity of the hands/arms) that prevents game playing as reported by the participant or observed by the Investigator.
4. Recent history (6 months prior to screening) of substance use disorder
5. History of seizures (excluding febrile seizures), significant tics, or a current diagnosis of Tourette's Disorder.
6. Known sensitivity to playing video games, such as photo-sensitive epilepsy, light-headedness, dizziness, nausea or motion sickness.
7. Participation in a clinical trial within 3 months prior to screening.
8. Plans to initiate, or to make significant changes in frequency, of non-pharmacological behavioral therapy during the study
9. Color blindness as detected by Ishihara Color Blindness Test
10. Urine test positive for nicotine or marijuana
11. Any other medical condition that in the opinion of the Investigator may confound study data/assessments.
12. Previous exposure to Akili Products within the 6 months prior to study enrollment
13. Plans to initiate or make significant changes to frequency or duration of non-pharmacological trainings with the aim to improve cognition by means of game or app-based cognitive trainings or neurofeedback, during the study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Primary objective of this study is to evaluate the efficacy of AKL-T01 as determined by the change in a digitally assessed measure after 4 weeks of treatment | After 4 weeks of treatment with AKL-T01
  Test of Variables of Attention (TOVA)-Attention Comparison Score (ACS) of sustained and selective attention. Measures at Day 1 and Exit/Post-Treatment Visit Day 28
  TOVA ACS is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. ACS is calculated using the following formula:
  ACS = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80 where Response Time is the average time it takes to respond correctly to a target, d' score is a response discriminability score reflecting the ratio of hits to "false alarms", and Variability is a measure of consistency of speed of responding based on the standard deviation of the mean correct response times. ACS tells how similar the score is to the ADHD profile. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.

SECONDARY OUTCOMES:
Secondary objective of this study is to evaluate the change in ADHD symptoms | After 4 weeks of treatment with AKL-T01
  Change in the Attention Deficit Hyperactive Disorder (ADHD) Rating Scale-5 inattention sub-scale and total scale scores. Measures taken at Baseline Visit (Day 1) and Exit/Post-Treatment Visit (Day 28).
  ADHD Rating Scale-5 is a clinician-administered questionnaire completed by the child's parent. The scale consists of two symptom subscales: Inattention and Hyperactivity-Impulsivity. The Inattention subscale raw score is computed by summing the item scores for 9 items. The total score is obtained by adding the Inattention and Hyperactivity-Impulsivity subscale raw scores. Each item is rated on a 4-point scale; Never or Rarely (0), Sometimes (1), Often (2), Very Often (3) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors.

OTHER OUTCOMES:
To evaluate the change in patient and caregiver perceived cognitive deficits | After 4 weeks of treatment with AKL-T01
  The change will be determined in selected items from the PROMIS® Parent Proxy Item Bank v1.1 - Cognitive Function and the PROMIS® Pediatric Item Bank v1.0-Cognitive Function
To evaluate changes in functional impairment | After 4 weeks of treatment with AKL-T01
  The change will be determined in ADHD-Rating Scale 5 Home Version relationship with significant others, peer relationships, academic functioning, behavioral functioning, homework functioning and self-esteem domains.
  ADHD Rating Scale-5 is a clinician-administered questionnaire completed by the child's parent. The scale asses six domains of impairment that are common among children with ADHD with one question item per domain. The scale is administered twice, once after each set of symptom subscale items (Inattention and Hyperactivity-Impulsivity). Each item is rated on a 4-point scale; No Problem (0), Minor Problem (1), Moderate Problem (2), Severe Problem (3). A higher score indicates more severe impairment due to ADHD symptoms and behaviors.
To evaluate changes in TOVA metrics other than ACS - Ex-Gaussian Tau Total | After 4 weeks of treatment with AKL-T01
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Ex-Gaussian Tau.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  * Ex-Gaussian Tau: The exponential decay (or "right hand tail") of the correct response times, modeled using the Ex-Gaussian distribution. Total refers to entire test (both H1 and H2). H1 refers to the first half of the test where target stimulus is infrequent (1 target to 3.5 non-targets), and H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate changes in TOVA metrics other than ACS - Commission Errors Standard Score H2 | After 4 weeks of treatment with AKL-T01
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Commission Errors Standard.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  -- Commission Errors Standard Score H2: Commission errors are the number of times the patient clicked the microswitch at the incorrect time. H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate changes in TOVA metrics other than ACS - Response Time Variability Standard Score Total | After 4 weeks of treatment with AKL-T01
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Response Time Variability Standard Score Total.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  - - Response Time Variability Standard Score Total: The standard score for the first standard deviation of the correct response times. Total refers to entire test (both H1 and H2). H1 refers to the first half of the test where target stimulus is infrequent (1 target to 3.5 non-targets), and H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate changes in TOVA metrics other than ACS - Response Time Mean Standard Score H1 | After 4 weeks of treatment with AKL-T01
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Response Time Mean Standard Score H1.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  * - Response Time Mean Standard Score H1:The standard score for the mean response time of the correct responses. H1 refers to the first half of the test where target stimulus is infrequent (1 target to 3.5 non-targets).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate changes in TOVA metrics other than ACS - D-Prime Standard Score H2 | After 4 weeks of treatment with AKL-T01
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - D-Prime Standard Score H2.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  -- D-Prime Standard Score H2: D-Prime score is a response discriminability score reflecting the ratio of hits to false alarms. The measure is derived from Signal Detection Theory and has been shown to help distinguish non-impaired individuals from those diagnosed with attention disorders. The score reflects the accuracy of target (signal) and nontarget (noise) discrimination and can be interpreted as a measure of perceptual sensitivity. H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate changes in TOVA metrics other than ACS - Omission Errors Standard Score H2 | After 4 weeks of treatment with AKL-T01
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Omission Errors Standard Score H2.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  - - Omission Errors Standard Score H2: Omission Errors are the number of times the patient failed to click the microswitch when the target was presented. H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate response rates for TOVA-ACS | After 4 weeks of treatment with AKL-T01
  The change will be determined in responder analyses for Test of Variables of Attention, Attention Comparison Score (TOVA-ACS).
  TOVA-ACS is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. ACS is calculated using a standardized formula.
  Responder rates will be 1.0-point improvement and TOVA-ACS greater then or equal to 1.0 at exit visit.
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.
To evaluate response rates for ADHD Rating Scale-5 | After 4 weeks of treatment with AKL-T01
  The change will be determined in responder analyses for ADHD Rating Scale 5.
  ADHD Rating Scale-5 is a clinician-administered questionnaire completed by the child's parent. The scale asses six domains of impairment that are common among children with ADHD with one question item per domain.
  Greater than or equal to 30% improvement in ADHD RS-5 total score from baseline after 4 weeks of AKL-T01 treatment.
  Measures at Day 1 and Exit/Post-Treatment Visit Day 28.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Melmed Center, Scottsdale, Arizona
  - Cortica, Inc., San Diego, California
  - Accel Research Sites, Maitland, Florida
  - MTP Psychiatry, Baltimore, Maryland
  - Midwest Research Group, Saint Charles, Missouri
  - Lincoln Pediatric Group, Lincoln, Nebraska
  - Alivation Research, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - MindPath Care Centers, Raleigh, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Southeast Houston Research, Inc., Houston, Texas

REFERENCES:
- [Derived] Stamatis CA, Heusser AC, Simon TJ, Ala'ilima T, Kollins SH. Real-time cognitive performance metrics derived from a digital therapeutic for inattention predict ADHD-related clinical outcomes: Replication across three independent trials of AKL-T01. Transl Psychiatry. 2024 Aug 11;14(1):328. doi: 10.1038/s41398-024-03045-0. PMID 39128918
- [Derived] Flannery JE, Hinshaw SP, Kollins SH, Stamatis CA. Secondary analyses of sex differences in attention improvements across three clinical trials of a digital therapeutic in children, adolescents, and adults with ADHD. BMC Public Health. 2024 Apr 29;24(1):1195. doi: 10.1186/s12889-024-18597-5. PMID 38685016